CLINICAL TRIAL: NCT04673305
Title: Cognitive Status Assessment In Elderly Patients With Active Treatment For Haematological Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale San Carlo Borromeo (Other)
Collaborators: Associazione Oncologica Milanese AmoLaVita ONLUS (Unknown)
Responsible Party: Principal Investigator, Vittorio Montefusco, Medical Director Ssd of Oncohaematology, Ospedale San Carlo Borromeo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Chemobrain Study
Record Dates: First submitted 2020-11-25; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cognitive Impairment; Haematological Malignancy; Chemo-brain
MeSH Terms: conditions — Cognitive Dysfunction; Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): patients ≥ 70 years, whith haematological malignancy, who need to start a treatment within 3 months
  Interventions: Other: Cognitive Assessment, Cytokine dosage

INTERVENTIONS:
Other: Cognitive Assessment, Cytokine dosage — Once the patient's informed consent has been acquired, a neurological examination is carried out, with functional tests required by the protocol. The patient carries out, as per clinical practice, the treatment provided for the cure of his disease. The evaluation of the tests is repeated at 6 months and 12 months after enrollment in the study. In conjunction with a venipuncture performed for the exams required by clinical management, a blood sample is taken to measure the cytokines involved in inflammatory processes.

SUMMARY:
BACKGROUND Neurocognitive symptoms have a high prevalence in cancer patients, resulting in a significant impact on daily life and tolerance to therapy. It's estimated that about 30% of cancer patients present a cognitive impairment before treatment, about 75% present this cognitive impairment during the treatment, and about 35% continue to present cognitive difficulties in the following months/years.

There is growing evidence that cognitive symptoms have a biological mechanism linked to the activation of immunological cytokines that exert important effects on the brain functions. For example, interferon α is known to increase the levels of IL-1, IL-6 and TNF-α, and this increase is associated with memory deficits, executive function and mood alterations.

A neurotoxic action induced by cytokines has been demonstrated both in the early stages of the tumor and after chemotherapy.

Several imaging studies suggest that the cognitive impairment pattern in cancer patients, during the treatment and in remission, is related to structural and functional brain changes.

Longitudinal studies in women with breast cancer treated with chemoterapy have shown a reduction in the volume of cerebral gray matter, mainly in the bilateral frontal cortex and hippocampus. In parallel, diffusion tensor imaging studies have shown an alteration of the integrity of the frontal, parietal and occipital cerebral white matter, demyelination and axonal degeneration processes. Finally, functional magnetic resonance studies in cancer patients have shown alterations in the connectivity of the default mode network compared to control subjects.

Studies carried out to date, show a prevalent impairment of executive functions and working memory. Cognitive impairment has been studied mainly as a possible adverse effect in women treated with chemotherapy for breast cancer, while there are few studies in the literature on patients with haematological malignancies.

STUDY DESIGN The study is targeted to patients ages ≥ 70 years, whith haematological malignancy, who need to start a treatment within 3 months.

Once the eligibility criteria have been assessed, the hematologist proposes the enrollment in the study. Once the patient's informed consent has been acquired, a neurological examination is carried out, functional tests required by the protocol are administered. The patient begins, as per clinical practice, the treatment provided for his/her haematological malignancy. Test's evaluation is repeated at 6 months and 12 months after the enrollment. In conjunction with neurological tests, will be performed a venipuncture as per clinical practice, and a blood sample is taken to measure the cytokines involved in inflammatory processes. It is expected that a patient can perform up to a maximum of 3 blood samples for the biological study.

STATISTICAL ANALYSIS This is a non-pharmacological, prospective, uncontrolled, open-label single-center interventional pilot study, aimed to describ the progress of cognitive function under treatment for haematological disease.

Due to the pilot and exploratory nature of the study and the substantial absence of a specific literature relating to the elderly onco-haematological patient, it is not believed that the conditions exist to be able to formally define the size of the sample. The sample size is arbitrarily fixed at 60 patients. The observation time will be 12 months from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥ 70 years;
* Signed Informed Consent Form;
* Haematological malignancy diagnosis that requires whithin three months a treatment.

Exclusion Criteria:

* Inability (ex. severe visual and/or hearing impairments, lack of caregivers) to carry out the tests required by the study;
* Comorbidity or condition that, in the investigator's opinion, may compromise the safe execution of the tests.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the score trend obtained with the Mini-mental test (MMSE) | 12 months from the enrollment
  MMSE score at 12 months will be compared with the MMSE at enrollment.

SECONDARY OUTCOMES:
Activities of daily living (ADL) score | 12 months from the enrollment
  ADL at 12 months will be compared with ADL at enrollment.
Instrumental activities of daily living (IADL) score | 12 months from the enrollment
  IADL at 12 months will be compared with IADL at enrollment.
Charlson comorbidity index | 12 months from the enrollment
  Charlson comorbidity index at 12 months will be compared with Charlson comorbidity index at enrollment.
CDT (clock drawing test) | 12 months from the enrollment
  CDT at 12 months will be compared with CDT st enrollment.
FAB (frontal assessment battery) | 12 months from the enrollment
  FAB at 12 months will be compared with FAB at enrollment.
Digit Span | 12 months from the enrollment
  Digit Span at 12 months will be compared with Digit Span at enrollment.
CorsiTest | 12 months from the enrollment
  Corsi Test at 12 months will be compared with Corsi Test at enrollment.
STAI-Y test | 12 months from the enrollment
  STAI-Y test at 12 months will be compared with STAI-Y test at enrollment.

OTHER OUTCOMES:
Serum IL-1 levels (pg/ml) | 12 months from the enrollment
  Correlations of IL-1 levels with cognitive functions.
Serum IL-2 levels (pg/ml) | 12 months from the enrollment
  Correlations of IL-2 levels with cognitive functions.
Serum IL-6 levels (pg/ml) | 12 months from the enrollment
  Correlations of IL-6 levels with cognitive functions.
Serum TNFα levels (pg/ml) | 12 months from the enrollment
  Correlations of TNFα levels with cognitive functions.
Serum IL-4 levels (pg/ml) | 12 months from the enrollment
  Correlations of IL-4 levels with cognitive functions.
Serum IL-10 levels (pg/ml) | 12 months from the enrollment
  Correlations of IL-10 levels with cognitive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Montefusco, MD, Principal Investigator — ASST SANTI PAOLO CARLO - SAN CARLO BORROMEO HOSPITAL; Fabio Frediani, MD, Principal Investigator — ASST SANTI PAOLO CARLO - SAN CARLO BORROMEO HOSPITAL
Locations (1):
- ASST SANTI PAOLO CARLO - SAN CARLO BORROMEO HOSPITAL - SSd. Onco - Haematology and SC Neurology, Milan, Italy

REFERENCES:
- [Background] Meyers CA, Albitar M, Estey E. Cognitive impairment, fatigue, and cytokine levels in patients with acute myelogenous leukemia or myelodysplastic syndrome. Cancer. 2005 Aug 15;104(4):788-93. doi: 10.1002/cncr.21234. PMID 15973668
- [Background] Pendergrass JC, Targum SD, Harrison JE. Cognitive Impairment Associated with Cancer: A Brief Review. Innov Clin Neurosci. 2018 Feb 1;15(1-2):36-44. PMID 29497579
- [Background] Ahles TA, Saykin AJ. Candidate mechanisms for chemotherapy-induced cognitive changes. Nat Rev Cancer. 2007 Mar;7(3):192-201. doi: 10.1038/nrc2073. PMID 17318212
- [Background] Ahles TA, Root JC, Ryan EL. Cancer- and cancer treatment-associated cognitive change: an update on the state of the science. J Clin Oncol. 2012 Oct 20;30(30):3675-86. doi: 10.1200/JCO.2012.43.0116. Epub 2012 Sep 24. PMID 23008308
- [Background] Deprez S, Amant F, Smeets A, Peeters R, Leemans A, Van Hecke W, Verhoeven JS, Christiaens MR, Vandenberghe J, Vandenbulcke M, Sunaert S. Longitudinal assessment of chemotherapy-induced structural changes in cerebral white matter and its correlation with impaired cognitive functioning. J Clin Oncol. 2012 Jan 20;30(3):274-81. doi: 10.1200/JCO.2011.36.8571. Epub 2011 Dec 19. PMID 22184379
- [Background] Deprez S, Billiet T, Sunaert S, Leemans A. Diffusion tensor MRI of chemotherapy-induced cognitive impairment in non-CNS cancer patients: a review. Brain Imaging Behav. 2013 Dec;7(4):409-35. doi: 10.1007/s11682-012-9220-1. PMID 23329357
- [Background] Simo M, Rifa-Ros X, Rodriguez-Fornells A, Bruna J. Chemobrain: a systematic review of structural and functional neuroimaging studies. Neurosci Biobehav Rev. 2013 Sep;37(8):1311-21. doi: 10.1016/j.neubiorev.2013.04.015. Epub 2013 May 6. PMID 23660455
- [Background] McDonald BC, Conroy SK, Ahles TA, West JD, Saykin AJ. Gray matter reduction associated with systemic chemotherapy for breast cancer: a prospective MRI study. Breast Cancer Res Treat. 2010 Oct;123(3):819-28. doi: 10.1007/s10549-010-1088-4. Epub 2010 Aug 6. PMID 20690040
- [Background] Hshieh TT, Jung WF, Grande LJ, Chen J, Stone RM, Soiffer RJ, Driver JA, Abel GA. Prevalence of Cognitive Impairment and Association With Survival Among Older Patients With Hematologic Cancers. JAMA Oncol. 2018 May 1;4(5):686-693. doi: 10.1001/jamaoncol.2017.5674. PMID 29494732
- [Background] Allegra A, Innao V, Basile G, Pugliese M, Allegra AG, Pulvirenti N, Musolino C. Post-chemotherapy cognitive impairment in hematological patients: current understanding of chemobrain in hematology. Expert Rev Hematol. 2020 Apr;13(4):393-404. doi: 10.1080/17474086.2020.1738213. Epub 2020 Mar 10. PMID 32129131
- [Background] Bradshaw M, Wefel J. The neuropsychology of oncology. In: Parsons M, Hammeke T (eds). Clinical Neuropsychology: A pocket handbook for assessment, Third edition. Washington DC: American Psychological Association; 2014:313-337